CLINICAL TRIAL: NCT00926159
Title: "Assessment of Appropriate ICD Implantation for Primary Prevention of Sudden Cardiac Death"
Brief Title: Assessment of Appropriate ICD Implantation for Primary Prevention of Sudden Cardiac Death
Status: Completed | Type: Observational
Sponsor: University of Minnesota Physicians Heart at Fairview (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Huagui Li, M.D., PhD, University of Minnesota Physicians
Other Study IDs: Version # 3, December 4, 2009
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-01

CONDITIONS: Cardiomyopathies
Keywords: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD eligible: Patients with Ejection Fraction (EF) of 35% or less as determined by cardiac echocardiogram or cardiac nuclear scan.

SUMMARY:
Prophylactic implant of an ICD (implantable cardioverter defibrillator) for prevention of sudden cardiac death from a life-threatening heart rhythm abnormality is a standard recommendation for patients with ejection fractions (EFs) of 35% or less. The main purpose of the trial is to determine why patients who are receiving care at a community-based cardiology program and are known to have a low ejection fraction (EF) measurement of 35% or less per echocardiogram and/or cardiac nuclear scan testing are not being approached for ICD (implantable cardioverter defibrillator) implant. Additionally, other secondary purposes of the trial are: 1) to determine if these patients are or are not receiving recommendation from their provider to undergo prophylactic ICD implant 2) identify the reasons providers are not recommending ICD implant for their patients with reduced EFs 3) determine reasons patients recommended for ICD implant by their provider elect not to have the implant.

DETAILED DESCRIPTION:
The implantable cardioverter defibrillator (ICD) for patients at high risk of sudden cardiac death (primary prevention) has become an accepted therapy after multiple randomized trials demonstrated the benefit consistently. After years of extensive evaluation of the trial data, Center for Medicare and Medicaid Services(CMS) has approved the national registry that is endorsed by the American College of Cardiology and Heart Rhythm Society. Thus, ICD implantation for primary prevention of sudden cardiac death is one of the most intensively evaluated, strictly regulated and closely monitored therapies.

Since the approval of expanded coverage for primary prevention by CMS along with the requirement for registry participation in early 2005, the ICD implant volume did not show an apparent increase as expected by many. Instead, a flat growth of ICD sales has been observed over the last 2 years. Several explanations have been offered by various sources. Some attribute the slow growth to the loss of confidence among the referring physicians, patients, and family members as the result of the multiple industry recalls. Others claim that only a small portion of the eligible candidates receive ICD therapy because of poor awareness of the ICD benefit among the referring physicians and the public (the Cambridge Heart Commercial). However, the Medtronic campaign to promote public awareness has had little impact on the volume of ICD implants. Another group of people suspect that the cardiologists have not paid enough attention to the patients' candidacy for ICD therapy because they tend to focus on the patients' ongoing symptoms not proactive prevention. Thus,an active screening program may identify a significant number of patients who will benefit from ICD therapy. However, there has been no comprehensive study that has evaluated the impact of active screening on the ICD implant volume, the percentage of eligible ICD patients without ICDs and the reasons for not receiving ICDs.

Majority of ICD implants in the United States are currently performed in the community-based cardiology programs. Thus a proactive program to identify ICD candidates in a community-based program may provide a good assessment on the unrealized potential benefit of ICDs for primary prevention of sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ejection fraction of 35% or less by echocardiogram and/or cardiac nuclear scan

Exclusion Criteria:

* Age less than 18 years
* Patients currently enrolled in a clinical trial that would be impacted by receipt of an ICD
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minnesota Heart Clinic Patients with an ejection fraction of 35% or less as identified from cardiac echocardiogram and/or cardiac nuclear scan.
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Minnesota Heart Clinic Provider progress note from the first office visit after the cardiac echocardiogram or nuclear scan that qualified the patient for inclusion in the trial will be reviewed for documentation of discussion regarding ICD implant. | First scheduled office visit with a Minnesota Heart Clinic Provider scheduled and conducted after the study qualifying cardiac echocardiogram or cardiac nuclear scan.

SECONDARY OUTCOMES:
A questionnaire will be issued/reviewed after completed by Providers to obtain reason(s) for not recommending ICD implant. | Questionnaire will be issued after review of progress note identifies no documentation regarding possible ICD implant.

CONTACTS AND LOCATIONS:
Overall Officials: Huagui Li, MD, PhD, Principal Investigator — University of Minnesota Physicians, Minnesota Heart Clinic